CLINICAL TRIAL: NCT06151561
Title: A Phase 1/2, Randomized, Double-Blinded, Placebo-Controlled Study of AGN-151586 in the Treatment of Japanese Subjects With Moderate to Severe Glabellar Lines
Brief Title: Study of AGN-151586 in Japanese Participants With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M24-040
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: Glabellar Lines, AGN-151586

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose 1 (Experimental): Participants will receive 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Dose 2 (Experimental): Participants will receive 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Dose 3 (Experimental): Participants will receive 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Placebo (Placebo Comparator): Participants will receive 5 intramuscular injections of Placebo in the glabellar complex on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular Injection
  Arms: Dose 1; Dose 2; Dose 3
Drug: Placebo — Intramuscular Injection
  Arms: Placebo

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to evaluate the safety and efficacy of AGN-151586 over a range of doses for the treatment of moderate to severe GL in Japanese participants.

AGN-151586 is an investigational product being developed for the treatment of GL. Participants are randomly assigned to receive AGN-151586 or placebo. There is 1 in a 4 chance that participants will receive placebo. Around 24 adult participants with moderate to severe GL will be enrolled in the study in approximately 2 sites in Japan.

Participants will receive either AGN-151586 or Placebo administered as 5 intramuscular injections to the glabellar complex on Day 1. The duration of the study will be approximately 6 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in good health as per investigator's judgment based on medical history, physical examination, neurological assessment, clinical laboratory evaluations, ECG results, and vital sign measurements.
* Participants must have moderate or severe GL at maximum frown as assessed by the investigator using the FWS-A at Screening and Baseline Day 1 Visit. The investigator ratings do not have to match between Screening and Baseline Day 1 Visit.

Exclusion Criteria:

* Participants must not have uncontrolled systemic disease.
* History of known immunization to any botulinum neurotoxin serotype
* Tattoos, jewelry, or clothing which obscure the glabellar area and cannot be removed.
* Anticipated need for surgery or overnight hospitalization during the study.
* History of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., rhinoplasty, facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* History of periorbital, mid-facial, or upper-facial treatment with semi permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Female subject who is pregnant or breastfeeding, and is considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
* Participant who has been treated with any investigational drug within 30 days of the drug prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* Anticipated need for treatment with botulinum neurotoxin of any serotype for any reason during the study (other than study drug).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a >= 2-grade improvement from baseline on the Facial Wrinkle Scale with Asian (FWS-A) Guide according to investigator assessment of Glabellar Lines (GL) severity at maximum frown, at any timepoint through Day 7 | Baseline (Day 1) through Day 7
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.

SECONDARY OUTCOMES:
Percentage of participants with a >= 2-grade improvement from baseline on the FWS-A according to investigator assessment of GL severity at maximum frown over time | Baseline (Day 1) through End of Study (Up to Day 42)
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of participants with a >= 1-grade improvement from baseline on the FWS-A according to investigator assessment of GL severity at maximum frown over time | Baseline (Day 1) through End of Study (Up to Day 42)
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of participants with a None or Mild on the FWS-A according to investigator assessment of GL severity at maximum frown over time | Baseline (Day 1) through End of Study (Up to Day 42)
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Tokyo Center Clinic /ID# 257898, Central District, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-040